CLINICAL TRIAL: NCT07290517
Title: The Carevix Device: Assessing Pain and Effectiveness of a Suction-based Cervical Stabilizer for IUD Insertions in the Clinic Setting: a Randomized, Controlled Trial (CARE)
Brief Title: Assessing Pain and Effectiveness of Carevix Device for IUD Insertions
Acronym: CARE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Aspivix SA (Industry)
Responsible Party: Principal Investigator, Alissa M Conklin, Assistant Professor of Clinical Obstetrics and Gynecology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 25731
Record Dates: First submitted 2025-12-11; First posted 2025-12-18 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-10

CONDITIONS: IUD; Abnormal Uterine Bleeding; Pain, Cervical
Keywords: IUD insertion; Cervical Stabilization; Tenaculum; Pain
MeSH Terms: conditions — Metrorrhagia; Neck Pain; Pain

STUDY DESIGN:
Masking Description: Patients will be randomized, but are unable to be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Carevix (Experimental): Patients will receive the atraumatic, suction-based, cervical stabilizer (Carevix) for their IUD insertion.
  Interventions: Device: Carevix
- Tenaculum (Active Comparator): Patients will receive the standard of care device (single tooth tenaculum) for their IUD insertion.
  Interventions: Device: Tenaculum

INTERVENTIONS:
Device: Carevix — Vacuum cervical stabilization device
  Arms: Carevix
Device: Tenaculum — Standard of care cervical stabilization device
  Arms: Tenaculum

SUMMARY:
The goal of this clinical trial is to evaluate patient-reported pain, bleeding, and device efficiency along with provider satisfaction and ease of use between IUD insertions using a suction cervical stabilizer (new device, FDA approved, atraumatic) and single-tooth tenaculum (standard, traumatic). Our aims are to:

* assess and compare patient-reported pain during IUD insertion between the Carevix device and tenaculum.
* assess predictors of pain scores including between nulliparous and multiparous patients
* assess provider-reported ease of use and satisfaction

Participants (including providers) will:

* be randomized to receive one device to complete the IUD procedure
* complete a survey following the procedure

DETAILED DESCRIPTION:
The primary objective is to assess and compare patient-reported pain during IUD insertion between the Carevix device and tenaculum. The hypothesis is that patient-reported pain scores comparing Carevix™ to tenaculum will be lower. The investigators will assess pain, and predictors for pain scores including nulliparous vs multiparous, when highest pain scores are reported, and expectation of pain for the procedure.

The secondary objective will be to assess Usability (provider assessment of ease of use, number of device placement attempts to secure sufficient traction on uterus), efficacy (ability to insert IUD with Carevix™ device alone without recourse to conventional tenaculum or other instruments), provider reported bleeding (cervical bleeding and ecchymosis), overall provider satisfaction, patient-reported pain scores at device placement prior to IUD insertion procedure and after completion of IUD insertion using Visual Analog Scale (VAS), overall patient satisfaction, and overall provider satisfaction. The investigators aim to expand the pilot trial data collection to assess cultural background, ethnicity and demographics while also assessing prior contraceptive choices, reasons for discontinuation of prior choices and reasons for current selection of IUD insertion and any anticipated barriers for removal.

ELIGIBILITY:
Inclusion Criteria (to be assessed prior to procedure):

* Age 18 years or older
* Able to consent on their own
* Scheduled and will undergo an IUD insertion within 90 days of consent
* Planned use of cervical stabilization device for placement
* Procedure being performed by a trained provider
* Provider is willing to use Carevix™ for scheduled procedure

Exclusion Criteria (to be assessed by provider at time of procedure):

* Vaginal bleeding of unknown origin
* Cervix less than 26 mm in diameter
* Nabothian cyst on anterior lip of cervix
* Cervical myomas
* Cervical abnormalities/shape
* Pregnant
* Participants who are not fluent in and/or do not fully understand, read, write, or speak the English language
* Other inability to provide informed consent to participate
* Initial attempt to place the IUD without any cervical stabilization

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Patient pain score (Numeric Pain Rating Scale) | During IUD insertion procedure
  0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"

SECONDARY OUTCOMES:
Provider device satisfaction | Immediately after IUD insertion procedure
  Questionnaire
Reason for IUD procedure | Immediately after IUD insertion procedure
  Questionnaire

OTHER OUTCOMES:
Predictors for pain score | Immediately after IUD insertion procedure
  Questionnaire
Patient pain score at device placement, prior to IUD insertion (Numeric Pain Rating Scale) | During IUD insertion procedure
  0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"
Patient pain score after completion of IUD insertion procedure (Numeric Pain Rating Scale) | Immediately after IUD insertion procedure
  0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"

CONTACTS AND LOCATIONS:
Overall Officials: Alissa M Conklin, MD, Principal Investigator — Indiana School of Medicine
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yaron M, Legardeur H, Barcellini B, Akhoundova F, Mathevet P. Safety and efficacy of a suction cervical stabilizer for intrauterine contraceptive device insertion: Results from a randomized, controlled study. Contraception. 2023 Jul;123:110004. doi: 10.1016/j.contraception.2023.110004. Epub 2023 Mar 11. PMID 36914147
- See also: Sponsor journal article — https://pubmed.ncbi.nlm.nih.gov/36914147/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-09-09): https://cdn.clinicaltrials.gov/large-docs/17/NCT07290517/Prot_SAP_000.pdf
  • Informed Consent Form (2025-09-25): https://cdn.clinicaltrials.gov/large-docs/17/NCT07290517/ICF_001.pdf